CLINICAL TRIAL: NCT00204165
Title: MRI of the Small Bowel. Comparison of Different Techniques and Contrast.
Brief Title: Comparison of MR Enteroclysis and MRI With Per Oral Contrast Using a 6 % Mannitol Solution.
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University of Oslo (Other)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Diagnostic
Other Study IDs: 431-04150
Record Dates: First submitted 2005-09-13; First posted 2005-09-20 (Estimated); Last update posted 2006-09-11 (Estimated); Status verified 2006-09

CONDITIONS: Magnetic Resonance Imaging, Intestine Small, Crohn Disease.
MeSH Terms: conditions — Crohn Disease

INTERVENTIONS:
Procedure: MRI of the small bowel

SUMMARY:
The purpose of this study is to compare MRI enteroclysis with MRI of the small bowel with a per oral 6%mannitol solution.Our hypothesis is that the peroral technique preform the same way as MRI Enteroclysis.

ELIGIBILITY:
Inclusion Criteria:

* above 18 years
* known Crohns disease or strong suspicion.
* need of a small bowel examination

Exclusion Criteria:

* pregnant
* electrolyte disturbances.
* Any MRI contraindications.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40
Dates: Start 2004-11; Study Completion 2005-06

CONTACTS AND LOCATIONS:
Overall Officials: Nils-Einar Kløw, Prof. MD, Study Director — Ulleval Universitetssykehus
Locations (1):
- Ulleval Universitets sykehus, Kirkeveien 166, Oslo County, Norway